CLINICAL TRIAL: NCT02338557
Title: Effectiveness of Motor Relearning Programme and Mirror Therapy Along With Conventional Physiotherapy Treatment for Improving Hand Function In Patients With Stroke.
Brief Title: Effect of Motor Relearning Programme and Mirror Therapy Along for Improving Hand Function In Patients With Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DIVYA MIDHA, EFFECTIVENESS OF MOTOR RELEARNING PROGRAMME AND MIRROR THERAPY ON HAND FUNCTIONS IN PATIENTS WITH STROKE., Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D789
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: STROKE
Keywords: MRP, MIRROR THERAPY, STROKE
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

ARMS (2):
- GROUP A (Experimental): Subjects in Group A received MRP exercises for training of Wrist Extensors, Extension of wrist and holding objects, training of supination of forearm, opposition of thumb, cupping of hand and training of manipulation of the objects.
  Interventions: Device: motor relearning programme
- GROUP B (Active Comparator): Group B received Mirror therapy in which patient was seated close to the table in front of mirror (35x35 cm). The involved hand was placed behind the mirror. : the practice consisted of intransitive exercises as Hand opening, Wrist extension and flexion, Forearm pronation and supination, Hand sliding on a flat surface. During the session patient were asked to try to do the same movement with the paretic hand while they were moving the non-paretic hand.In both the groups total treatment was given for 1 hour/day for 6 days/week
  Interventions: Device: MIRROR THERAPY

INTERVENTIONS:
Device: motor relearning programme — MRP exercises for training of Wrist Extensors, Extension of wrist and holding objects, training of supination of forearm, opposition of thumb, cupping of hand and training of manipulation of the objects
  Other Names: MRP
  Arms: GROUP A
Device: MIRROR THERAPY — Mirror therapy in which patient was seated close to the table in front of mirror (35x35 cm). The involved hand was placed behind the mirror. : the practice consisted of intransitive exercises as Hand opening, Wrist extension and flexion, Forearm pronation and supination, Hand sliding on a flat surface. During the session patient were asked to try to do the same movement with the paretic hand while they were moving the non-paretic hand.In both the groups total treatment was given for 1 hour/day for 6 days/week
  Arms: GROUP B

SUMMARY:
Study was conducted Effectiveness of Motor Relearning Programme and Mirror Therapy along with Conventional Physiotherapy treatment for improving Hand Function In Patients with stroke. study was an experimental study conducted on 12 stroke patients using convenient sampling method .Subjects were divided into two equal groups (n=6). Group A was given conventional physiotherapy and Motor Relearning Programme exercises for the affected hand and Group B received conventional physiotherapy for the affected hand and mirror therapy for the unaffected hand. Chedoke arm and hand inventory (CAHAI) was used as primary outcome measure for evaluation of hand function before and after application of therapeutic Intervention

DETAILED DESCRIPTION:
Title: Effectiveness of Motor Relearning Programme and Mirror Therapy along with Conventional Physiotherapy treatment for improving Hand Function In Patients with stroke.

Background Upper extremity complications are common following stroke. Individuals who have sustained stroke are often left with residual motor deficits of the upper limb. These deficits restrict functional use of the limb in everyday activities and can result in increased dependen cy upon others to engage in some tasks.

Objectives Present study aims to see effectiveness of mirror therapy and Motor Relearning Programme for improving hand functions in stroke.

Materials and Methods Present study was an experimental study conducted on 12 stroke patients using convenient sampling method .Subjects were divided into two equal groups (n=6). Group A was given conventional physiotherapy and Motor Relearning Programme exercises for the affected hand and Group B received conventional physiotherapy for the affected hand and mirror therapy for the unaffected hand. Chedoke arm and hand inventory (CAHAI) was used as primary outcome measure for evaluation of hand function before and after application of therapeutic Intervention

ELIGIBILITY:
Inclusion Criteria:

* experienced one episode of stroke only,
* Both ischemic & hemorrhagic stroke individuals
* Duration of stroke between 1 to 6 months,
* Mini mental status examination (MMSE) (score > 23),
* Brunstrom Stage 4 & 5.

Exclusion Criteria:

* any musculoskeletal Disorders,
* neurological disorder other than stroke,
* visual impairment, systemic disease,
* Non co-operative patients
* psychological problems.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Chedoke arm and hand activity inventory (CAHAI) | 4 WEEKS
  CAHAI scale is designed to encourage the bilateral hand to complete the task. Patient was made to seat in chair without arm rest and encouraging erect posture with elbows at the edge of the table and hands resting on the table. Each task was demonstrated once before performance, and then the Score was evaluated of the affected upper extremity using the 7 point activity scale from total assistance (1) to complete independence.

SECONDARY OUTCOMES:
MODIFIED ASHWSORTH SCALE | 4 WEEKS
  to assess the level of spasticity